CLINICAL TRIAL: NCT06077409
Title: ''The Effect of Skin-to-Skin Contact and Gentle Touch Method Applied During Blood Collection on Early Detection of Pain and Physiological Parameters''
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, DERYA KILINÇ, Assisstant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 177
Record Dates: First submitted 2023-09-21; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Venipuncture; Pain; Touch
Keywords: pain; pretem; physiological findings; gentle human touch; skin to skin; touch
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Premature babies who apply to the blood collection room to take blood, were included in the gentle human touch, skin to skin and control groups. Randomization occurred on: www.randomizer.org
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gentle Human Touch Group (Active Comparator): After the mother is dressed in a clean apron, she will be provided to wash and disinfect her hands and heat her hand temperature with a non-contact fire meter device until the measurement value is 34 ºC.Jul. The mother, who was previously informed about the method, will place the fingertips and palm of one hand above the eyebrow line so that it touches the baby's crown part, while placing the other hand on the lower abdomen surrounding the baby's waist and hips (Figure 1). The GHT application will be started 5 minutes before the blood collection procedure, it will be continued during the blood collection procedure and until 5 minutes after the end of the blood collection procedure.
  Interventions: Behavioral: Gentle Human Touch
- Skin to Skin Group (Active Comparator): The temperature of the environment where skin to skin will be carried out will be adjusted between 22-26 degrees C. The mother will be allowed to disinfect her hands and warm them until her hand temperature is at least 34 C. Only the baby's diaper, hat and socks will be left behind, and the baby will be placed face down on the mother's chest, with its head upright and its legs under the breasts in a frog position. The baby's face will be turned towards the mother and eye contact will be made. The baby will be in an upright position between the mother's breasts and skin to skin with the mother.
  Skin-to-skin contact will begin 5 minutes before blood collection, continue throughout the procedure, and skin to skin will continue until 5 minutes after the procedure.
  Interventions: Other: Skin To Skin
- Control Group (No Intervention): The standard procedure of the clinic was applied to preterm infants in the control group. In the standart prosedure of the clinic, the mother was with her baby in the blood collection room and did not perform any procedure.

INTERVENTIONS:
Other: Skin To Skin — Skin to Skin Contact Group The temperature of the environment where kangaroo care will be carried out will be adjusted between 22-26 degrees C. The mother will be allowed to disinfect her hands and warm them until her hand temperature is at least 34 C. Only the baby's diaper, hat and socks will be left behind, and the baby will be placed face down on the mother's chest, with its head upright and its legs under the breasts in a frog position. The baby's face will be turned towards the mother and eye contact will be made. The baby will be in an upright position between the mother's breasts and skin to skin with the mother.
  Skin-to-skin contact will begin 5 minutes before blood collection, continue throughout the procedure, and kangaroo care will continue until 5 minutes after the procedure.
  Arms: Skin to Skin Group
Behavioral: Gentle Human Touch — Experimental Group (Gentle Touch/Gentle Human Touch-GHT); After the mother is dressed in a clean apron, her hands are washed and disinfected, and it is safe to warm the hand temperature with a non-contact thermometer device until the measured value is 34 ºC. The mother, who was previously informed about the method, will be placed on the eyebrow line with the crown piece that will separate the fingertips and tuft of one hand, while the other hand will be placed on the lower abdomen, which will mark the waist and hips (Figure 1). The blood collection amount of GHT application will be started 5 minutes before, make sure that the blood collection is done and the blood collection will continue until 5 minutes later.
  Arms: Gentle Human Touch Group

SUMMARY:
37. babies under the gestational week are considered preterm babies, and babies between 32-37 gestational weeks are considered late preterm babies (WHO, 2023). Dec. While the preterm birth rate in the world is 10%, this rate is 13% in Turkey. The life rate of preterm babies has increased in recent years and they are subjected to many painful interventions for diagnosis, treatment and preventive purposes. At the time of birth, they experience painful interventions such as vitamin K, hepatitis B vaccine administration, heel blood collection. Painful interventions cause an increase in cortisol levels, resulting in impaired blood sugar in infants, impaired brain development, impaired growth and development (Akyildiz et al., 2023). In the short term, they may give signs of a decrease in oxygen saturation, an increase in heart rate, metabolic acidosis( Akcan et al., 2017). Procedural pain management is also important for the neurological development of preterm infants (Perg et al., 2018). For these reasons, the pain of the newborn due to interventional procedures should be managed well.

DETAILED DESCRIPTION:
Newborns are often exposed to acute or chronic pain due to different invasive interventions (Akcan and Polat, 2017). The American Pain Society (APS) accepts pain as the fifth physiological parameter (McCharty et al., 2013). The American Academy of Pediatrics (AAP) recommends minimizing pain due to invasive procedures (Aydın et al., 2016). Reducing pain first requires accurate assessment of pain and treatment with pharmacological/non-pharmacological interventions (Hussein, 2015). Pharmacological methods have risks such as drug-related side effects. For this reason, non-pharmacological methods are primarily preferred in acute pain (Hashemi et al., 2016).

Non-pharmacological methods for pain management are diverse. In recent years, non-pharmacological methods such as distraction, wrapping, positioning, aromatherapy, music, games, massage, kangaroo care, and oral sucrose have been used together or separately to reduce pain and/or stress-related behaviors (Abdallah et al., 2013).

In another application, the tent-to-skin contact method, the newborn is laid face down on the parent's chest. The newborn's back is covered to prevent heat loss. It is thought that this situation will relax the newborn and therefore perceive the pain as milder (Mayfield, 2019).

Gentle Human Touch is one of the therapeutic touch methods. Gentle touch, which is a simple and applicable method in newborns, is a non-invasive touch technique that does not require special equipment and technology. The gentle touch method is a sensitive tactile stimulation applied to the skin, without caressing or massage, and provides a relaxing effect on the baby (Dur et al., 2020; Fatohallazade, 2020).

Newborns need their parents, especially their mothers, to be with them during all kinds of interventions. For this reason, the parent should be with the newborn during the invasive interventions and take a primary role in the non-pharmacological interventions; It provides optimum comfort for the nurse, newborn and caregiver. It is important to benefit from the family-centered care model when using non-pharmacological methods. Family-centered care is a care model based on collaboration between health professionals and children's families in the planning, delivery and evaluation of health services. Its general goal is to increase the quality of health services for children and families, increase the satisfaction of families and health professionals, and ensure the effective use of personnel (Yılmaz and Gözen, 2019).

It was planned as a randomized controlled experimental design type in order to determine the importance of the family-centered care model and parents' participation in the procedures and to determine the effect of non-pharmacological methods applied to preterm newborns by their mothers on the pain occurring during blood collection and the effect on preterm physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who volunteer to participate in the research,
* Between 32-37 weeks of gestation,
* No analgesics are given until 6 hours before the procedure,
* First blood draw attempt is successful,
* Those who are considered healthy by the physician in the health follow-ups performed after birth

Exclusion Criteria:

* Those with congenital anomalies,
* Having any disease,
* Patients whose intravenous blood collection attempt takes more than two minutes,
* Babies previously monitored in the Neonatal Intensive Care Unit will be excluded from the scope of the research.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Preterm Pain | 5 minutes. At the first mınute of venipuncture Scores will be given between 0-7 points.
  Neonatal İnfant Pain Scale
Preterm Crying | 5 mınutes. During blood collection, the stopwatch will turn on when the baby starts crying and turn off when the baby stops crying.
  Stopwatch

SECONDARY OUTCOMES:
Heart Rate | 1.Five minutes before the blood collection procedure, 2. In the first minute of the blood collection process 3. Five minutes after the blood collection procedure
  Measured 3 times in total
Oxygen Saturatıon | 1.Five minutes before the blood collection procedure, 2. In the first minute of the blood collection process 3. Five minutes after the blood collection procedure
  Measured 3 times in total

CONTACTS AND LOCATIONS:
Overall Officials: Derya Kılınç, 1, Principal Investigator — Istanbul Cerrahpaşa
Locations (1):
- Istanbul Provincial Health Directorate Zeynep Kamil Women and Children Diseases Traning and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdallah B, Badr LK, Hawwari M. The efficacy of massage on short and long term outcomes in preterm infants. Infant Behav Dev. 2013 Dec;36(4):662-9. doi: 10.1016/j.infbeh.2013.06.009. Epub 2013 Aug 7. PMID 23932956
- [Background] Aydin D, Sahiner NC, Ciftci EK. Comparison of the effectiveness of three different methods in decreasing pain during venipuncture in children: ball squeezing, balloon inflating and distraction cards. J Clin Nurs. 2016 Aug;25(15-16):2328-35. doi: 10.1111/jocn.13321. Epub 2016 Apr 26. PMID 27112434
- [Background] Ayyildiz TK, Tanriverdi E, Tank DY, Akkoc B, Topan A. The effect of swaddling method applied to preterm infants during the aspiration procedure on pain. J Pediatr Nurs. 2023 May-Jun;70:61-67. doi: 10.1016/j.pedn.2022.05.025. Epub 2023 Feb 18. PMID 36801626
- [Background] Baley J; COMMITTEE ON FETUS AND NEWBORN. Skin-to-Skin Care for Term and Preterm Infants in the Neonatal ICU. Pediatrics. 2015 Sep;136(3):596-9. doi: 10.1542/peds.2015-2335. PMID 26324876
- [Background] Dur S, Caglar S, Yildiz NU, Dogan P, Guney Varal I. The effect of Yakson and Gentle Human Touch methods on pain and physiological parameters in preterm infants during heel lancing. Intensive Crit Care Nurs. 2020 Dec;61:102886. doi: 10.1016/j.iccn.2020.102886. Epub 2020 Jun 27. PMID 32601011
- [Background] Fatollahzade M, Parvizi S, Kashaki M, Haghani H, Alinejad-Naeini M. The effect of gentle human touch during endotracheal suctioning on procedural pain response in preterm infant admitted to neonatal intensive care units: a randomized controlled crossover study. J Matern Fetal Neonatal Med. 2022 Apr;35(7):1370-1376. doi: 10.1080/14767058.2020.1755649. Epub 2020 Apr 21. PMID 32316790
- [Background] Hashemi F, Taheri L, Ghodsbin F, Pishva N, Vossoughi M. Comparing the effect of swaddling and breastfeeding and their combined effect on the pain induced by BCG vaccination in infants referring to Motahari Hospital, Jahrom, 2010-2011. Appl Nurs Res. 2016 Feb;29:217-21. doi: 10.1016/j.apnr.2015.05.013. Epub 2015 May 30. PMID 26856517
- [Background] McCarthy M, Glick R, Green J, Plummer K, Peters K, Johnsey L, Deluca C. Comfort First: an evaluation of a procedural pain management programme for children with cancer. Psychooncology. 2013 Apr;22(4):775-82. doi: 10.1002/pon.3061. Epub 2012 Mar 13. PMID 22416039
- [Background] Pavlyshyn H, Sarapuk I. Skin-to-skin contact-An effective intervention on pain and stress reduction in preterm infants. Front Pediatr. 2023 Mar 22;11:1148946. doi: 10.3389/fped.2023.1148946. eCollection 2023. PMID 37033163
- [Background] Peng HF, Yin T, Yang L, Wang C, Chang YC, Jeng MJ, Liaw JJ. Non-nutritive sucking, oral breast milk, and facilitated tucking relieve preterm infant pain during heel-stick procedures: A prospective, randomized controlled trial. Int J Nurs Stud. 2018 Jan;77:162-170. doi: 10.1016/j.ijnurstu.2017.10.001. Epub 2017 Oct 8. PMID 29100198
- See also: Akcan, E. & Polat, S. (2017). Yenidoğanlarda Ağrı ve Ağrı Yönetiminde Hemşirenin Rolü. Acıbadem Üniversitesi Sağlık Bilimleri Dergisi, (2): 64-69 — http://journal.acibadem.edu.tr/tr/download/article-file/1701610
- See also: Mayfield, A. (2019). Effects of Kangaroo Mother Care on Mother-Infant Interaction: Infant Behaviors (Doctoral dissertation, Southeast Missouri State University). — https://www.proquest.com/docview/2300291088?pq-origsite=gscholar&fromopenview=true
- See also: WHO Preterm Birth Detail — http://www.who.int/news-room/fact-sheets/detail/preterm-birth
- See also: Yılmaz, Ö. E., & Gözen, D. (2019). Pediatri Hemşireliğinde Aile Merkezli Bakımın Önemi ve Bakım Kalitesini Geliştirmedeki Değeri. Türkiye Klinikleri Çocuk Sağlığı ve Hastalıkları Hemşireliği-Özel Konular, 5(2), 5-11. — http://www.turkiyeklinikleri.com/journal/cocuk-sagligi-ve-hastaliklari-hemsireligi-ozel-konular/461/issue/2019/5/2-0/pediatri-hemsireliginde-aile-merkezli-bakim/tr-index.html